CLINICAL TRIAL: NCT00912197
Title: Effect of Oligofructose on Appetite, Gut Hormones and Body Composition in Healthy Overweight Subjects
Brief Title: Effect of Oligofructose on Appetite in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CRO1243
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Appetite Regulation; Obesity
Keywords: Appetite regulation; Oligofructose intake
MeSH Terms: conditions — Obesity | interventions — oligofructose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligofructose (Experimental): Participants received 10g of Oligofructose powdered supplements in sachets each containing 10 g dietary fiber) three times per day. Volunteers were instructed to take the supplement with their main meals.The 8-week supplementation period took place between visits 3 and 4 and included a 2-week run-in period to allow the bowel to adapt to the 30 g of dietary fiber.
  Interventions: Dietary Supplement: Oligofructose
- Cellulose and maltodextrin (Placebo Comparator): Participants received 10g of Cellulose powdered supplements in sachets each containing 10 g dietary fiber) three times per day. Volunteers were instructed to take the supplement with their main meals. Maltodextrin was added to the cellulose supplement. The 8-week supplementation period took place between visits 3 and 4 and included a 2-week run-in period to allow the bowel to adapt to the 30 g of dietary fiber.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligofructose — Participants will be asked to consume 30g of oligofructose daily for six weeks after a 2-week run-in.
  Arms: Oligofructose
Dietary Supplement: Placebo — Participants will be asked to consume 3 doses (a total of 30g dietary fibres) of the placebo product daily for six weeks after a 2-week run-in
  Arms: Cellulose and maltodextrin

SUMMARY:
This study seeks to look into the effects of oligofructose supplementation on appetite, energy intake, and body weight and body composition in overweight subjects. Compared to a placebo product (cellulose) oligofructose is hypothesised to suppress hunger and thereby reduce food intake moderately leading to a decrease in body weight.

DETAILED DESCRIPTION:
Appetite regulation plays an important part in energy balance. Suppressing appetite by manipulating the diet is a safe way of reducing energy intake and body weight compared to drug therapy and obesity surgery. How various nutrients affect appetite is not fully understood. Non-digestible carbohydrates (NDC) may affect appetite differently due to differences in physio-chemical properties.

This project will look into how two different NDC affect appetite and energy intake in overweight individuals in a randomised, double-blinded, placebo controlled parallel study. The NDC under investigation are oligofructose and cellulose, both natural compounds of plant origin. The former is broken down (fermented) in the large bowel by friendly bacteria producing various compounds that may affect appetite and the metabolism of the host.

Volunteers will consume one of the two NDC for eight weeks (including a two week run-in period). Appetite study session, functional MRI (fMRI) and MRI body fat scans will be conducted before and after the supplementation with NDC (or during the supplementation in the case of fMRI). Using fMRI the effect of the NDC supplementation on central appetite regulating centres will be investigated. Appetite questionnaires and dietary records will completed under free-living conditions at baseline and during the supplementation to explore the effect on subjective appetite feelings and energy intake, respectively.

It is hoped that this project will enhance the understanding of how NDC affect appetite and provide further information on how fermentation of NDC, gut hormone release, body composition, and appetite regulation are linked.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 20-50
* BMI 25-35 kg/m2
* Weight stable for three months prior to enrollment in study (weight change < 3 kg over a period of three months)
* Habitual dietary fibre ≤ 25g/day (as assessed by 3-day dietary record)
* Non-smokers
* No current or history of endocrine disease, gastrointestinal disease, kidney or liver diseases, cardiovascular disease, pancreatitis, or cancer
* Hydrogen producers

Exclusion Criteria:

* Use of antibiotic less than three months prior to participation in the study
* Participation in other research studies in the previous three months
* Blood donation less than three months before participation in study
* Anaemia
* Hypertension
* Pregnancy or breastfeeding
* Substance abuse
* Vegan diet
* Regular use of prebiotic, probiotic or symbiotic food items/ supplements
* Intense exercise undertaken for more than 5h per week
* Metallic or electronic implants e.g. pacemaker, cochlear ear implants, fixed dental braces
* Claustrophobia
* Depression

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Frost, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pedersen C, Lefevre S, Peters V, Patterson M, Ghatei MA, Morgan LM, Frost GS. Gut hormone release and appetite regulation in healthy non-obese participants following oligofructose intake. A dose-escalation study. Appetite. 2013 Jul;66:44-53. doi: 10.1016/j.appet.2013.02.017. Epub 2013 Mar 5. PMID 23474087
- [Result] Daud NM, Ismail NA, Thomas EL, Fitzpatrick JA, Bell JD, Swann JR, Costabile A, Childs CE, Pedersen C, Goldstone AP, Frost GS. The impact of oligofructose on stimulation of gut hormones, appetite regulation and adiposity. Obesity (Silver Spring). 2014 Jun;22(6):1430-8. doi: 10.1002/oby.20754. Epub 2014 Apr 8. PMID 24715424

RESULTS

PARTICIPANT FLOW:
Groups:
- Oligofructose: Participants consumed 30g of oligofructose daily for 6 weeks after a 2-weeks run-in.
- Cellulose and Maltodextrin: Placebo: Participants consumed 3 doses (a total of 30g dietary fibres) product daily for six weeks after a 2-week run-in
Period: Overall Study
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Started | 15 | 13
Completed | 12 | 10
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oligofructose | Cellulose and Maltodextrin | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (2.2) | 28.7 (2.3) | 32 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 10 | 22
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (1.0) | 31.1 (1.1) | 30.5 (1.1)
waist:hip ratio (WHR) [Mean (Standard Deviation); unit: ratio] | 0.86 (0.03) | 0.82 (0.02) | 0.84 (0.02)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Appetite Ratings in Hunger Compared to Baseline
Description: Hunger was assessed by visual analogue scales (Each scale is 10cm in length with words anchored at each end, expressing the most positive (Minimum score = 0 cm and means no hunger) and the most negative rating (Maximum score = 10 cm and means very hungry). Compared to baseline after treatment at 56 days
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: cm
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
cm
  baseline | 4.8 (0.9) | 3.6 (0.8)
  56 days | 3.6 (0.8) | 4.1 (0.6)
Statistical Analysis 1: Comparison: Oligofructose vs Cellulose and Maltodextrin; Test type: Superiority; p = 0.135, ANCOVA

2. Primary Outcome: Subjective Appetite Ratings in Fullness Compared to Baseline
Description: Fullness are assessed by visual analogue scale, 10 cm in length with words anchored at each end, expressing the most positive (feel full: maximum Score=10cm) and the most negative rating (feeling empty: Minimum Score = 0cm), values at baseline and after treatments at 56 days
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
units on a scale
  Baseline | 4.7 (0.5) | 4.2 (0.8)
  56 days | 4.2 (0.8) | 4.1 (0.6)
Statistical Analysis 1: Comparison: Oligofructose vs Cellulose and Maltodextrin; Test type: Superiority; p = 0.688, ANCOVA

3. Primary Outcome: Body Weight
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: kg
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
kg
  Baseline | 83.7 (4.9) | 86 (4.4)
  56 days | 84.1 (4.8) | 86.3 (4.5)
Statistical Analysis 1: Comparison: Oligofructose vs Cellulose and Maltodextrin; after treatment, 56 days; Test type: Superiority; p = 0.715, t-test, 2 sided

4. Primary Outcome: Energy Intake
Description: Energy intake was assessed by 7-days food diary at baseline and last week of treatment, diaries were analysed by Dietplan6 software.
  The values in the table represent the Energy intake as measured over the whole week (as opposed to reporting the Energy intake per day based on the 7 day data).
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: kcal
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
kcal
  Baseline | 873.16 (54.06) | 867.61 (159.45)
  56 days | 760.19 (51.59) | 725.34 (117.40)
Statistical Analysis 1: Comparison: Oligofructose vs Cellulose and Maltodextrin; Test type: Superiority; p = 0.578, ANCOVA
Statistical Analysis 2: Comparison: Oligofructose; baseline to after treatment, at 56 days; Test type: Superiority; p = 0.007, t-test, 2 sided
Statistical Analysis 3: Comparison: Cellulose and Maltodextrin; baseline to after treatment, at 56 days; Test type: Superiority; p = 0.05, t-test, 2 sided — calculated

5. Primary Outcome: Gut Hormone PYY
Description: Total PYY concentrations were quantified using specific and sensitive in-house radio-immunoassays as previously described.
Time Frame: baseline (Day 0) and post-supplementation (Day 56)
Population: The PI has left the institution. There is no access to the raw data, we only have access to the graphical data in publication (please see: Daud NM, Ismail NA, Thomas EL, Fitzpatrick JA, Bell JD, Swann JR, Costabile A, Childs CE, Pedersen C, Goldstone AP, Frost GS. The impact of oligofructose on stimulation of gut hormones, appetite regulation and adiposity. Obesity (Silver Spring). 2014 Jun;22(6):1430-8. doi: 10.1002/oby.20754. Epub 2014 Apr 8. PubMed ID: 24715424 for graph)
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Body Composition
Description: Body composition assessed by BMI
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
kg/m^2
  Baseline | 29.7 (1.0) | 31.1 (1.1)
  56 days | 29.9 (1.1) | 31.2 (1.1)

7. Secondary Outcome: Imaging of Total Adipose Tissue
Description: Total adipose tissue was assessed by FMRI at baseline and after treatment period
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: percentage of body fat
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
percentage of body fat
  Baseline | 36.3 (2.8) | 38.4 (3.7)
  56 days | 37 (2.8) | 38.7 (3.8)

8. Secondary Outcome: Plasma Short-chain Fatty Acids Concentrations After Treatment
Description: Short-chain fatty acids (acetate, propionate, butyrate) concentrations assessed from plasma at 56 days at 450min timepoint with gas chromatography
Time Frame: Baseline, 56 days
Measure: Mean (Standard Error); unit: uM
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
uM
  Acetate | 81.3 (2.1) | 72.8 (1.8)
  Propionate | 5.4 (0.6) | 5.4 (0.6)
  Butyrate | 0.9 (0.1) | 0.7 (0.2)
Statistical Analysis 1: Comparison: Oligofructose vs Cellulose and Maltodextrin; Acetate; Test type: Superiority; p = 0.024, ANCOVA

9. Secondary Outcome: Inflammatory Markers
Description: No data were collected for this Outcome Measure
Time Frame: baseline (Day 0) and post-supplementation (Day 56)
Population: Inflammatory markers where never measured for this study and so therefore no results available.
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Glycemic Response
Description: Glucose was analyzed in the Department of Clinical Biochemistry, Hammer-smith Hospital, London using an Abbott Architect ci8200 analyzer(Abbott Diagnostics, Maidenhead, UK).
Time Frame: baseline (Day 0) and post-supplementation (Day 56)
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
mmol/L | 4.8 [4.6 to 5.0] | 4.7 [4.5 to 5.0]

11. Secondary Outcome: Serum Insulin
Description: Plasma insulin concentrations were assayed using RIA kits (Millipore, MO).
Time Frame: baseline (Day 0) and post-supplementation (Day 56)
Measure: Mean (95% Confidence Interval); unit: (mU/L
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 12 | 10
(mU/L | 10.2 [8.7 to 12] | 9.6 [6.4 to 15.6]

12. Secondary Outcome: Breath Hydrogen Levels
Description: breath hydrogen were obtained from volunteers throughout the study session.
Time Frame: baseline (Day 0) and post-supplementation (Day 56)
Population: as for outcome 5
Arm/Group | Oligofructose | Cellulose and Maltodextrin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Oligofructose | Cellulose and Maltodextrin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes